CLINICAL TRIAL: NCT06714136
Title: The Role of miRNA in Group 3 Pulmonary Hypertension
Acronym: miRNA-GR3PH
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: miRNA-GR3PH; RC22000410 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2024-11-28; First posted 2024-12-03 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Lung tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PAH (idiopathic pulmonary hypertension): Patients with idiopathic pulmonary hypertension
- IPF-PH (idiopathic pulmonary fibrosis and pulmonary hypertension): Patients with idiopathic pulmonary fibrosis and pulmonary hypertension
- COPD-PH (COPD and pulmonary hypertension): Patients with COPD and pulmonary hypertension

SUMMARY:
This study recognizes the substantial value of lung tissue obtained from explanted lungs for fundamental research purposes.By analyzing pulmonary tissue affected by pulmonary hypertension, it is possible to discover shared pathogenetic mechanisms between these two groups and to gain a deeper understanding of the mechanisms underlying pulmonary hypertension.

DETAILED DESCRIPTION:
Lung transplantation serves as the sole therapeutic approach targeting the enhancement of life expectancy and quality of life for individuals afflicted with advanced parenchymal or vascular lung diseases. The current study aligns with this objective, recognizing the substantial value of lung tissue obtained from explanted lungs for fundamental research purposes. By investigating lung tissue affected by both group 3 and group 1 pulmonary hypertension, it becomes possible to uncover shared pathogenic mechanisms between these two groups and gain a more profound understanding of the underlying mechanisms driving group 3 pulmonary hypertension. Furthermore, delving into the cells responsible for the expression of dysregulated miRNAs offers the potential to identify novel target mechanisms for the clinical management of group 3 pulmonary hypertension, an area currently limited in therapeutic options. Through a comparative analysis of the quantitative expression patterns of each miRNA among distinct groups, it becomes feasible to determine the extent of involvement of specific pathogenic pathways in the various forms of pulmonary hypertension. Consequently, this approach provides guidance for future research, directing focus towards the most relevant mechanisms of interest.

ELIGIBILITY:
Inclusion criteria

* Patients who underwent lung transplantation at the AOU IRCCS Policlinico Sant'Orsola in Bologna and the IRCCS Fondazione Policlinico San Matteo in Pavia (satellite center) from January 1, 2010, to December 31, 2021.
* Diagnosis of idiopathic pulmonary arterial hypertension, idiopathic pulmonary fibrosis, or chronic obstructive pulmonary disease.
* Patients who underwent at least one pre-transplant right heart catheterization in clinically stable conditions, with findings of mPAP ≥ 25 mmHg, PVR > 3 WU, and PCP < 15 mmHg.
* Suitability of lung explant tissue available in the archives of the participating pathology departments: presence of at least 3 pulmonary arterioles in each specimen.
* Acquisition of informed consent. Exclusion criteria
* Unsuitability of lung tissue for molecular biology investigations (due to preservation issues or deterioration of the necessary arteriolar structures).
* Patients with active neoplastic diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tissue samples from lung explants of patients who underwent lung transplantation at IRCCS University Hospital of Bologna and at IRCCS San Matteo Hospital of Pavia from the 1st of January 2010 to the 31th of December 2021 were considered. Among 149 transplant performed in the two transplant center during the period of interest, we included in this study 27 patients who were submitted to single or double lung transplant with the following indications: idiopathic pulmonary arterial hypertension and idiopathic pulmonary fibrosis, or chronic obstructive pulmonary disease, both complicated by pulmonary arterial hypertension (defined as PAPm ≥ 25 mmHg) All patients underwent right heart catheterization during pre-transplant screening and had explanted lung samples available for the study.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
miRNAs espression | 18 months
  expression of miRNAs underlying the development of pulmonary arterial hypertension shared between idiopathic pulmonary arterial hypertension and pulmonary arterial hypertension in patients with idiopathic pulmonary fibrosis and chronic obstructive pulmonary disease.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Salvaterra, MD, PhD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS AOU Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No